CLINICAL TRIAL: NCT01850901
Title: Renal Sympathetic Denervation as a New Treatment for Therapy Resistant Hypertension - A Multicenter Randomized Controlled Trial
Brief Title: Renal Sympathetic Denervation as a New Treatment for Therapy Resistant Hypertension
Acronym: SYMPATHY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Medtronic (Industry)
Responsible Party: Principal Investigator, P. J. Blankestijn, Peter J. Blankestijn, nephrologist, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-540
Record Dates: First submitted 2013-03-21; First posted 2013-05-10 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hypertension; Chronic Kidney Disease
Keywords: Hypertension; Renal denervation; Sympathetic denervation
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Renal sympathetic denervation (Experimental): Catheter-based renal nerve ablation
  Interventions: Procedure: Renal sympathetic denervation
- Usual care (No Intervention): Antihypertensive treatment according to guidelines

INTERVENTIONS:
Procedure: Renal sympathetic denervation
  Arms: Renal sympathetic denervation

SUMMARY:
The aim of this study is to assess whether renal denervation (RD) added to usual care compared to usual care alone reduces blood pressure (BP) as determined with ambulatory BP monitoring (ABPM) after 6 months in subjects with an average day-time systolic BP of at least 135 mmHg as determined with use of ABPM, despite use of three or more BP lowering agents or with documented intolerance or contraindication for to 2 or more of the 4 major classes of antihypertensive drugs (ACEi/ARB, calcium channel blockers, betablockers and diuretics) obstructing use of 3 antihypertensives

Further aims are to assess the effect of renal denervation on the use of BP lowering agents, to explore the effect of renal denervation in strata of estimated glomerular filtration rate (eGFR) (eGFR 20-60 mL/min per 1.73m2 and eGFR>60 mL/min per 1.73m2) and according to baseline office BP.

Randomization will be stratified by hospital and eGFR and will be at a 2:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. Individual has a mean day-time SBP ≥ 135 mmHg, as determined with the use of ABPM, while using 3 or more antihypertensive agents for at least 3 months prior to inclusion or with documented intolerance to 2 or more of the 4 major classes antihypertensive drugs ( ACE/ARB, Calcium channel blocker, Beta Blocker, Diuretic) and no possibility to take 3 anti-hypertensive drugs.
2. Individual is ≥18 years of age.

Exclusion Criteria:

1. Individual is unable or unwilling to sign informed consent.
2. Individual has a treatable secondary cause of hypertension.
3. Individual has an eGFR below 20 mL/min/1.73m2 using the Modification of Diet in Renal Disease (MDRD) calculation.
4. Individual has renal artery anatomy that is ineligible for treatment
5. Individual has any serious medical condition, which in the opinion of the investigator, may adversely affect the safety and/or effectiveness of the participant or the study.
6. Individual is pregnant, nursing or planning to be pregnant.
7. Individual has a known, unresolved history of drug use or alcohol dependency, lacks the ability to comprehend or follow instructions, or would be unlikely or unable to comply with study follow-up requirements.
8. Individual is currently enrolled in another investigational drug or device trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2013-05; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in BP (measured by ABPM) | 6 months
  Change in BP: average day-time systolic blood pressure (SBP) as determined with the use of ambulatory blood pressure-monitoring at 6 months and during prolonged follow up (total 2 years)

SECONDARY OUTCOMES:
Change in the amount of antihypertensive medication | 6 months
  Change in antihypertensive medication defined as daily defined dose (DDD) of all prescribed drugs after 6 months and during prolonged follow up (total: 2 years)
Change in BP in eGFR strata | 6 months
  The effect on BP of RD in strata of eGFR: eGFR 20-60 mL/min per 1.73m2 versus eGFR>60 mL/min per 1.73m2 at 6 months after intervention and during prolonged follow up (total 2 years)
Change in office BP | 6 months
  Change in office blood pressure at 6 months after intervention and during follow up (total 2 years)

OTHER OUTCOMES:
Impact on quality of life | 6 months
  Impact on quality of life of RD will be measured with Short-Form 36 and EuroQol-5 Dimensions (EQ-5D) measurement instruments. Assessments at 6 months and during prolonged follow up (total 2 years)
Cost-effectiveness | 6 months
  Cost-effectiveness of RD will be calculated. For this purpose, health care and indirect costs will be monitored with use of data from the case report form and questionnaires. Absence from work will be assessed using parts of the Short-Form Health and Labour Questionnaire. Assessments at 6 months and during prolonged follow up (total 2 years)

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] de Jager RL, de Beus E, Beeftink MM, Sanders MF, Vonken EJ, Voskuil M, van Maarseveen EM, Bots ML, Blankestijn PJ; SYMPATHY Investigators. Impact of Medication Adherence on the Effect of Renal Denervation: The SYMPATHY Trial. Hypertension. 2017 Apr;69(4):678-684. doi: 10.1161/HYPERTENSIONAHA.116.08818. PMID 28264922
- [Derived] Vink EE, de Beus E, de Jager RL, Voskuil M, Spiering W, Vonken EJ, de Wit GA, Roes KC, Bots ML, Blankestijn PJ. The effect of renal denervation added to standard pharmacologic treatment versus standard pharmacologic treatment alone in patients with resistant hypertension: rationale and design of the SYMPATHY trial. Am Heart J. 2014 Mar;167(3):308-314.e3. doi: 10.1016/j.ahj.2013.11.010. Epub 2013 Dec 4. PMID 24576513